CLINICAL TRIAL: NCT01661803
Title: Intrathecal Bupivacaine Versus Bupivacaine and Clonidine in Paediatrics Age Group:A Comparative Evaluation
Status: Completed | Type: Observational
Sponsor: ACPM Medical College (Other)
Responsible Party: Principal Investigator, DR.NAGESH JAMBURE, resident,anesthesia department,a.c.p.m.medical college,dhule,maharashtra,india, ACPM Medical College
Other Study IDs: acpm anesthesia.dhule.
Record Dates: First submitted 2012-08-04; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Pediatric Spinal Anesthesia
Keywords: bupivacaine; clonidine; pediatric spinal; efficacy; duration; quality; side effects; intrathecal bupivacaine alone; bupivacaine plus clonidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group-A and group-B: Group-A (0.5% hyperbaric bupivacaine 0.4 mg/kg for 5-15 kg or 0.3mg/kg for >15kg) and Group-B (0.5% hyperbaric bupivacaine 0.4 mg/kg for 5-15 kg or 0.3mg/kg for >15 with 1 mcg/kg preservative free clonidine).
- group-A and group--B: Group-A (0.5% hyperbaric bupivacaine 0.4 mg/kg for 5-15 kg or 0.3mg/kg for >15kg) and Group-B (0.5% hyperbaric bupivacaine 0.4 mg/kg for 5-15 kg or 0.3mg/kg for >15 with 1 mcg/kg preservative free clonidine).

SUMMARY:
The investigators can summarize intrathecal clonidine can potentiate bupivacaine thereby bringing about better quality and longer duration of analgesia, better sedation and better postoperative outcomes with minimal side effects.

DETAILED DESCRIPTION:
In our Randomized controlled, double blind study involving 30 subjects in two groups; the investigators compared the safety, efficacy and quality of using intrathecal hyperbaric bupivacaine 0.5% and hyperbaric bupivacaine 0.5% with clonidine 1µg/kg in paediatric patients undergoing surgeries below T8 dermatome.

American Society of Anesthesiologists (ASA) Grade I patients aged between 3-10 years were scheduled for the surgeries below T8 dermatome up to two hrs duration. The patients were randomly allocated in - Group A-who received 0.5%of hyperbaric Bupivacaine 0.4mg/kg for 5 to15 kg or 0.3 mg/kg for more than 15 kg intrathecally.

Group B-who received 0.5%of hyperbaric Bupivacaine 0.4mg/kg for 5 to15 kg or 0.3 mg/kg for more than 15 kg and 1µg/kg preservative free clonidine intrathecally.

The patients studied across the group did not vary much with respect to age, weight and sex distribution.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade-1 physical status.
2. weight 5-35kg
3. age-3 to 10 yrs

Exclusion Criteria:

1. patients with known sensitivity to drugs to be used.
2. gross spinal deformity
3. patients in whom regional anesthesia is contraindicated.
4. patients with peripheral neuropathy.
5. patient with hemodynamic instability.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: prospective,randomized,double blind study cariied in 60 ASA grade 1 pediatric patients undergoing surgeries below T8 dermatome upto two hours duration.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)